CLINICAL TRIAL: NCT07203131
Title: Evaluation of the Impact of an Alteration of NAD+ Metabolism on the Renal Prognosis of Patients Admitted to Intensive Care
Brief Title: Evaluation of the Impact of an Alteration of NAD+ Metabolism on the Renal Prognosis of Patients Admitted to Intensive Care (NI-AKI)
Acronym: NI-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-A01709-36
Record Dates: First submitted 2025-05-26; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Renal Insufficiency; NAD
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient admitted to intensive care for a high-risk reason of ARI (Experimental): Patient admitted to intensive care for a high-risk reason of ARI : Shock, Sepsis, Cardiovascular arrest, Post-operative unscheduled surgery, Post-operative cardiac surgery
  Interventions: Diagnostic Test: Urine sample; Other: Phone call at day 28

INTERVENTIONS:
Diagnostic Test: Urine sample — 5 mL of urine when the patient is admitted in intensive care To look for possible acute renal failure in the patient
Other: Phone call at day 28 — It will allow the following information to be collected:
  * Post-resuscitation monitoring and length of hospitalization,
  * Vital status,
  * Collection of adverse events,
  * Concomitant treatments.

SUMMARY:
Among all patients admitted to intensive care, it is estimated that more than half of them are exposed during their stay to acute renal failure (ARF). Impacting the vital prognosis to short term, the occurrence of renal failure is not without consequences in intensive care survivors, presenting an increased risk of death mainly mediated by an excess risk with regard to chronic kidney disease and/or certain cardiovascular pathologies.

Malnutrition, particularly vitamin deficiency, has already been reported as a risk factor for AKI. Studies on two models (animal and human) have recently highlighted the importance of NAD+ production failure in the onset of renal failure.

NAD+ synthesis can be done from tryptophan or via a salvage pathway from vitamin PP.

In a phase 2 study in patients undergoing cardiac surgery, vitamin B3 supplementation was accompanied by a reduction in the occurrence of AKI and a limitation of the duration / intensity of renal dysfunction.

This innovative research aims to identify an alteration in the metabolic pathway of NAD+ production as a risk factor for AKI in intensive care patients. This would be the first study to address this issue in this specific population.

The main objective of this research is to describe the association between the urinary Quinolinate/Tryptophan ratio on admission and the occurrence of acute renal failure in patients admitted to intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female aged over 18,
* Patient admitted to intensive care for a reason with a high risk of ARI: shock, sepsis, cardio-circulatory arrest, post-operative unscheduled surgery, post-operative cardiac surgery,
* Patient with normal renal function on admission,
* Patient affiliated to or beneficiary of a social security scheme,
* Patient having been informed and having given his/her free, informed and written consent

Exclusion Criteria:

* Minor patient,
* History of chronic kidney disease,
* History of kidney transplant,
* Admission for a reason with a low risk of ARI (neuroresuscitation, voluntary drug intoxication with anxiolytics - antidepressants - psychotropic drugs),
* Acute non-infectious respiratory failure, (scheduled surgery other than cardiac surgery)
* Patient hospitalized without consent,
* Patient in a period of exclusion due to another research still in progress at the time of inclusion,
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision,
* Pregnant, breastfeeding or parturient woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Acute renal insufficiency | 2 days
  * An increase in creatinine ≥ 0.3 mg/dL (26.5 μmol/L) within 48 hours
  * Or an increase in creatinine ≥ 1.5 times the baseline value
  * Or a urine volume < 0.5 mL/kg/h over a 6-hour period
  * Urinary Quinolinate/Tryptophan (Q/T) ratio on admission

SECONDARY OUTCOMES:
ARI Features : severity of ARI | 12 hours
  * grad 1 : creatinine between 1.5 and 1.9 times the baseline value OR increase ≥ 0.3 mg/dL (26.5 μmol/l) and urine < 0.5 mL/kg/h over a period of 6h to 12h
  * grad 2 : creatinine between 2.0 and 2.9 times the base value and urine < 0.5 mL/kg/h over a duration ≥12
  * grad 3 : creatinine greater than or equal to 3.0 times the baseline value OR increase ≥ 4.0 mg/dL (353.6 μmol/L) OR use of extra-renal purification OR patients under 18 years of age with decrease in creatinine clearance < 35 mL/min per 1.73 m² and urine < 0.3 mL/kg/h over a duration of ≥24h OR anuria over a duration of ≥12h
Duration or ARI | between 1 day and 28 days
  Duration in days of ARI
Cardiovascular complications | between day 1 and day 7
  * evolution of the troponin level between D1 and D7,
  * Use of mechanical ventilation and duration,
  * Evolution of the SOFA score between D1 and D7
Patient follow-up | 28 days
  Mortality within 28 days of admission to intensive care, NI-AKI
  * Number of days alive outside intensive care within 28 days of admission to intensive care,
  * Number of days alive not hospitalized within 28 days of admission to intensive care.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de l'Ouest Parisien, Trappes, France

IPD SHARING:
Plan to Share IPD: No